CLINICAL TRIAL: NCT00000548
Title: Inhaled NO in Prevention of Chronic Lung Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Prevention
Other Study IDs: 92; U01HL062514 (NIH)
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Bronchopulmonary Dysplasia; Lung Diseases
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Lung Diseases | interventions — Respiration, Artificial

INTERVENTIONS:
Procedure: mechanical ventilation

SUMMARY:
To test the hypothesis that low-dose inhaled nitric oxide administered to preterm infants who continue to require mechanical ventilation at 14 days of age will reduce the incidence of chronic lung disease.

DETAILED DESCRIPTION:
BACKGROUND:

Respiratory morbidity, particularly chronic lung disease (CLD), remains a major cause of long-term morbidity and mortality for preterm infants. Although surfactant replacement has decreased acute respiratory morbidity and mortality, it has not reduced the incidence of CLD. A number of other approaches, including antenatal thyrotropin releasing hormone in conjunction with corticosteroids, postnatal steroid administration, as well as administration of Vitamin E, diuretics, and bronchodilators, have not resulted in clinically important decreases in CLD. Infants with the most severe CLD go on to develop findings suggestive of pulmonary hypertension with cor pulmonale. There is preliminary evidence in the preterm infant with severe chronic lung disease that low-dose inhaled nitric oxide may significantly attenuate the disease and decrease mortality.

DESIGN NARRATIVE:

The multi-center, controlled and blinded trial investigates the hypothesis that low-dose inhaled nitric oxide administered to preterm infants between 500 and 1250 grams birth weight who continue to require mechanical ventilation at 10 days of age will increase survival without chronic lung disease (CLD) at 36 weeks post menstrual age. Secondary outcomes are duration of ventilation, oxygen requirement and duration of hospitalization. In addition, that there will be expected improvement in infant respiratory status (ventilatory support, airway resistance and compliance) associated with inhaled nitric oxide treatment. Indicators of inflammation and oxidant stress will be assessed by measurements of specific cytokines and protein modifications in tracheal aspirate and plasma samples, respectively. The safety of this therapy will be evaluated by assessing toxicity as measured by clinical bleeding, including intraventricular hemorrhage as well as the incidence of other morbidities of the preterm infant (necrotizing enterocolitis, retinopathy of prematurity and infection) and assessing neurodevelopmental outcome through two years of age. A total of 480 infants were randomized to either inhaled NO or placebo. In summary, this clinical trial will assess the efficacy and safety of inhaled nitric oxide for amelioration of a major disease of premature infants.

ELIGIBILITY:
Preterm infants who are 500-1250 grams at birth and who require mechanical ventilation at 10 to 21 days of age. Exclusions include congenital heart disease or pulmonary abnormalities, including a patent ductus arteriosus, ventilation solely for apnea, small-for-gestational age, or clinical bleeding.

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 2000-03; Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Survival without chronic lung disease (CLD) | 36 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Roberta Ballard — Children's Hospital of Philadelphia

REFERENCES:
- [Background] Ballard PL, Merrill JD, Godinez RI, Godinez MH, Truog WE, Ballard RA. Surfactant protein profile of pulmonary surfactant in premature infants. Am J Respir Crit Care Med. 2003 Nov 1;168(9):1123-8. doi: 10.1164/rccm.200304-479OC. Epub 2003 Aug 6. PMID 12904326
- [Background] Merrill JD, Ballard RA, Cnaan A, Hibbs AM, Godinez RI, Godinez MH, Truog WE, Ballard PL. Dysfunction of pulmonary surfactant in chronically ventilated premature infants. Pediatr Res. 2004 Dec;56(6):918-26. doi: 10.1203/01.PDR.0000145565.45490.D9. Epub 2004 Oct 20. PMID 15496605
- [Derived] Walsh MC, Hibbs AM, Martin CR, Cnaan A, Keller RL, Vittinghoff E, Martin RJ, Truog WE, Ballard PL, Zadell A, Wadlinger SR, Coburn CE, Ballard RA; NO CLD Study Group. Two-year neurodevelopmental outcomes of ventilated preterm infants treated with inhaled nitric oxide. J Pediatr. 2010 Apr;156(4):556-61.e1. doi: 10.1016/j.jpeds.2009.10.011. Epub 2010 Feb 6. PMID 20138299
- [Derived] Zupancic JA, Hibbs AM, Palermo L, Truog WE, Cnaan A, Black DM, Ballard PL, Wadlinger SR, Ballard RA; NO CLD Trial Group. Economic evaluation of inhaled nitric oxide in preterm infants undergoing mechanical ventilation. Pediatrics. 2009 Nov;124(5):1325-32. doi: 10.1542/peds.2008-3214. Epub 2009 Oct 19. PMID 19841125
- [Derived] Ballard RA, Truog WE, Cnaan A, Martin RJ, Ballard PL, Merrill JD, Walsh MC, Durand DJ, Mayock DE, Eichenwald EC, Null DR, Hudak ML, Puri AR, Golombek SG, Courtney SE, Stewart DL, Welty SE, Phibbs RH, Hibbs AM, Luan X, Wadlinger SR, Asselin JM, Coburn CE; NO CLD Study Group. Inhaled nitric oxide in preterm infants undergoing mechanical ventilation. N Engl J Med. 2006 Jul 27;355(4):343-53. doi: 10.1056/NEJMoa061088. PMID 16870913